CLINICAL TRIAL: NCT01378299
Title: CYP19A1 Gene and Pharmacogenetics of Response
Brief Title: CYP19A1 (Cytochrome P450 Family 19 Subfamily A Member 1) Gene and Pharmacogenetics of Response to Testosterone Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: SPLC-001-10S
Record Dates: First submitted 2011-06-16; First posted 2011-06-22 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Hypogonadism
Keywords: testosterone
MeSH Terms: conditions — Hypogonadism | interventions — testosterone 17 beta-cypionate; Testosterone Propionate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1: Testosterone Cypionate (Experimental): All patients who qualify for the study will receive testosterone cypionate
  Interventions: Drug: Testosterone Cypionate

INTERVENTIONS:
Drug: Testosterone Cypionate — Testosterone cypionate was administered at 200 mg by intramuscular injection every 2 weeks.
  DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Testosterone cypionate is a white or creamy white crystalline powder, odorless or nearly so and stable in air. It is insoluble in water, freely soluble in alcohol, chloroform, dioxane, ether, and soluble in vegetable oils. The chemical name for testosterone cypionate is androst-4-en-3-one,17-(3-cyclopentyl-1oxopropoxy)-, (178)-. Its molecular formula is CvH400a, and the molecular weight of 412.61.
  Other Names: depo testosterone

SUMMARY:
Testosterone (T) replacement prevents bone loss and relieves symptoms associated with androgen deficiency in male patients with hypogonadism, but at the expense of an increase in prostate-related adverse events and in the hematocrit values above the normal which may lead to bad circulatory outcomes. Most of the effects of T on the male skeleton are mediated by its conversion to estradiol (E2) by the enzyme aromatase. Genetic variations in the aromatase (CYP19A1) gene result in enzymes with variable activity and variable levels of E2 and T. This project is designed to determine if genetic variations in the CYP19A1 gene will result in differences in the skeletal response and incidence of side effects from T treatment in patients with low T. A large number of male Veterans are on T. Results from this project will help identify patients who would benefit from the therapy from those at risk for side effects, and would definitely have an impact in the future care of these patients and male patients in general once genetic profiling becomes part of the standard of care.

DETAILED DESCRIPTION:
Estrogen has been gaining recognition as the primary hormone that regulates the male skeleton. Estrogen in males is mainly derived from the conversion of testosterone to estradiol by the enzyme aromatase. Polymorphisms of the aromatase gene (CYP19A1) have been reported to result in variable enzyme activity resulting in variable hormonal profile and differences in bone mineral density (BMD) among the variants. These polymorphisms were also found to influence changes in BMD in response to hormone therapy in postmenopausal women and bone loss from aromatase inhibitors in women with breast cancer. It is possible that these same polymorphisms will also influence skeletal response to testosterone therapy in hypogonadal males given testosterone.

Among the side effects described for testosterone therapy, prostate-related events and an increase in hematocrit represent as the more common and the potentially more serious side effects. However, these side effects do not affect everybody, suggesting that a certain subgroup of patients is predisposed to these side effects. Because polymorphisms in the CYP19A1 gene result differences in activity among variants leading in variable substrate and product accumulation, the investigators hypothesize that these polymorphisms will influence the skeletal response and perhaps susceptibility to side effects from testosterone therapy. Thus the objectives of this proposal are: (1) To evaluate the influence of polymorphisms in the CYP19A1 gene on the skeletal response to testosterone in male patients with low testosterone, (2) To evaluate the influence of polymorphisms in the CYP19A1 gene on the susceptibility to side effects from testosterone therapy, (3) To evaluate the changes in functional activity of the aromatase enzyme in clinically significant CYP19A1 gene polymorphisms. The investigators propose to treat 105 patients with testosterone cypionate 200 mg IM every 2 weeks for an 18-month treatment period. The investigators will do serial measurements of BMD by dual energy X-ray absorptiometry, markers of bone turnover, hematocrit, prostate-specific antigen (PSA), prostate volume and hormonal assays. Changes in BMD and markers of bone turnover with testosterone treatment will be compared among the different CYP19A1 genotypes. The investigators will also compare changes in hematocrit, PSA and prostate volume among the different CYP19A1 genotypes. Changes in functional activity among the variants will be evaluated by CYP19 gene expression studies on the adipose tissues obtained from periumbilical fat biopsies, and by changes the in estradiol to testosterone ratio, a surrogate marker for aromatase activity. The investigators anticipate that variants with increase in activity will have relatively higher estradiol levels than less active variants resulting in greater increments in BMD. Meanwhile, less active variants will have relatively higher levels of testosterone than other variants and have greater increments in hematocrit. On the other hand, variants associated with higher estradiol to testosterone ratio will experience greater increases in PSA and prostate volume with therapy.

The incidence of testosterone deficiency goes up with aging and the presence of co-morbid conditions making male hypogonadism one of the common problems among patients attending the VA clinics who, are for the most part, elderly with various co-morbid conditions. Indeed, a large number of VA patients are already taking testosterone for hypogonadism, some of them primarily to prevent further bone loss. It is possible that some of these patients do not derive benefit from the drug while subjecting them to potential serious side effects. Results from this proposal will identify the genetic profiles of favorable responders from poor responders or those who might be more prone to serious side effects, thus, may impact the future care of male Veterans and hypogonadal patients in general, once genetic profiling becomes part of the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Male Veterans with low total testosterone (<300 ng/dl) as defined by the Endocrine Society, who are between 40-75 years of age.
* These patients must be ambulatory; and be willing and able to provide written informed consent.

Exclusion Criteria:

* history of prostate cancer, breast cancer
* history of testicular disease
* untreated sleep apnea
* any ongoing illness that, in the opinion of the investigator, could prevent the subject from completing the study
* patients with a hematocrit of more than 50% (2010 Endocrine Society Guidelines)
* prostate-related findings of a palpable prostate nodule on exam, a serum PSA of 4.0 ng/ml or more, International Prostate Symptom Score >8(9), urinary postvoid residual by ultrasound of >149 ml, or an abnormal transrectal ultrasound
* patients who are on androgen replacement therapy, selective androgen receptor modulator, or finasteride
* patients currently on medications that affects bone metabolism such as:

  * estrogen
  * the selective estrogen receptor modulator (SERM) as raloxifene
  * use of bisphosphonates (i.e. risedronate, alendronate, zoledronic acid and pamidronate)
  * within two years of study entry
  * aromatase inhibitors
  * GnRH analogs
  * glucocorticoids of at least 5 mg daily for one month or more
  * anabolic steroids
  * dilantin
  * warfarin
* patients with diseases known to interfere with bone metabolism as hyperparathyroidism, untreated hyperthyroidism, osteomalacia, chronic liver disease, renal failure, hypercortisolism, malabsorption and immobilization
* those with current alcohol use of more than 3 drinks per day (62).
* history of documented coronary artery disease at high risk for recurrence
* Subjects with osteoporosis or a BMD T-score of -2.5 in the lumbar spine, total femur or femoral neck as well as those patients with a history of osteoporosis-related fractures (spine, hip or wrist) or vertebral deformities on lateral spine radiographs deemed as fragility fractures by the team principal investigator.
* history of documented coronary artery disease at high risk for recurrence, history of deep vein thrombosis and cerebrovascular event.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male Veterans with low total testosterone (<300 ng/dl) as defined by the Endocrine Society, who are between 40-75 years of age.
Enrollment: 105 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2016-11-07 (Actual); Study Completion 2017-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reina C Villareal, MD, Principal Investigator — New Mexico VA Health Care System, Albuquerque, NM
Locations (2):
- United States (2):
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
People who ensure quality from the institutions where the research is being done, federal and other regulatory agencies will have access to all of the research data such as Food and Drug Administration (FDA) and Data Monitoring Committee (DMC). The purpose of collecting information covered under 38 U.S.C. 7332 is to conduct scientific research and no personnel involved in this study will identify, directly or indirectly, any individual patient or subject in any report of such research.
  The only research data that will leave the MEDVA MC will be emailed to the FDA and Data Monitoring Committee, and will include only data on subjects who developed side effects including heart attacks, strokes, high hematocrit, high PSA, psychiatric problems and other adverse events, and the results of their tests. None of the 18 HIPAA identifiers will be included.

REFERENCES:
- [Derived] Joad S, Ballato E, Deepika F, Gregori G, Fleires-Gutierrez AL, Colleluori G, Aguirre L, Chen R, Russo V, Fuenmayor Lopez VC, Qualls C, Villareal DT, Armamento-Villareal R. Hemoglobin A1c Threshold for Reduction in Bone Turnover in Men With Type 2 Diabetes Mellitus. Front Endocrinol (Lausanne). 2021 Dec 28;12:788107. doi: 10.3389/fendo.2021.788107. eCollection 2021. PMID 35027909
- [Derived] Colleluori G, Aguirre L, Napoli N, Qualls C, Villareal DT, Armamento-Villareal R. Testosterone Therapy Effects on Bone Mass and Turnover in Hypogonadal Men with Type 2 Diabetes. J Clin Endocrinol Metab. 2021 Jul 13;106(8):e3058-e3068. doi: 10.1210/clinem/dgab181. PMID 33735389

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Testosterone Cypionate: All patients who qualify for the study will receive testosterone cypionate
  Testosterone Cypionate: DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Subjects were divided into different groups of BMI.
  Testosterone cypionate is a white or creamy white crystalline powder, odorless or nearly so and stable in air. It is insoluble in water, freely soluble in alcohol, chloroform, dioxane, ether, and soluble in vegetable oils. The chemical name for testosterone cypionate is androst-4-en-3-one,17-(3-cyclopentyl-1oxopropoxy)-, (178)-. Its molecular formula is CvH400a, and the molecular weight 412.61.is available in two strengths, 100 mg/mL and 200 mg/mL testosterone cypionate.
Period: Overall Study
Arm/Group | Arm 1: Testosterone Cypionate
Started | 105
BMI group1 (BMI of <30 kg/m^2) | 38
BMI Group 2 (BMI between 30 to <35 kg/m^2) | 40
BMI Group 3 (BMI = or >35 kg/m^2) | 27
Completed | 74
Not Completed | 31

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Testosterone Cypionate: All patients who qualify for the study will receive testosterone cypionate
  Testosterone Cypionate: DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Subjects were divided into different groups of BMI.
  Testosterone cypionate is a white or creamy white crystalline powder, odorless or nearly so and stable in air. It is insoluble in water, freely soluble in alcohol, chloroform, dioxane, ether, and soluble in vegetable oils. The chemical name for testosterone cypionate is androst-4-en-3-one,17-(3-cyclopentyl-1oxopropoxy)-,
  (178)-. Its molecular formula is CvH400a, and the mole
Arm/Group | Arm 1: Testosterone Cypionate
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: years]
  BMI group 1 | 61.7 (8.5)
  BMI group 2 | 57.3 (8.7)
  BMI group 3 | 60.0 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants were divided into BMI groups.
  Participants
    BMI group 1: number analyzed (Participants) | 38
    BMI group 1: Female | 0
    BMI group 1: Male | 38
    BMI group 2: number analyzed (Participants) | 40
    BMI group 2: Female | 0
    BMI group 2: Male | 40
    BMI group 3: number analyzed (Participants) | 27
    BMI group 3: Female | 0
    BMI group 3: Male | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasians | 45
  Blacks | 11
  Hispanics | 33
  Asian | 1
  American Indian | 1
  Not reported | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 105
Body mass index [Mean (Standard Deviation); unit: kg/m2]
  BMI group 1 | 27.2 (1.9)
  BMI group 2 | 32.1 (1.4)
  BMI group 3 | 39.8 (3.9)
patients with diabetes mellitus [Count of Participants; unit: Participants]
  patients with diabetes mellitus | 49
  patients without diabetes mellitus | 56
aromatase activity as assessed using estradiol to testosterone ratio [Mean (Standard Deviation); unit: estradiol to testosterone ratio] — Aromatase activity was assessed using estradiol to testosterone ratio and the whole groups was divided equally according to tertiles of estradiol to testosterone ratio. Population: Only the first 87 participants analyzed for this assessment
  estradiol to testosterone ratio
    Tertile 1: number analyzed (Participants) | 29
    Tertile 1 | 0.069 (0.04)
    Tertile 2: number analyzed (Participants) | 29
    Tertile 2 | 0.25 (0.07)
    Tertile 3: number analyzed (Participants) | 29
    Tertile 3 | 1.37 (1.12)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Bone Mineral Density (BMD) According to rs700518 Polymorphism in the CYP19A1 Gene
Description: Percent change in bone mineral density from baseline to 18 months
Time Frame: form baseline to 18 months
Population: Analysis was by intention to treat with the last value carry forward. Those who had at least one follow-up from baseline were included in the analysis. The data from 84 subjects were available for analysis; 15 in the GG, 44 in the GA and 25 in the AA genotype.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- GG Genotype for RS 700518 Polymorphism of the CYP19A1 Gene: All patients who qualify for the study will receive testosterone cypionate
  Testosterone Cypionate: DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Subjects were divided into the different genotypes for the rs700518 polymorphism of the CYP19A1 gene.
  Testosterone cypionate is a white or creamy white crystalline powder, odorless or nearly so and stable in air. It is insoluble in water, freely soluble in alcohol, chloroform, dioxane, ether, and soluble in vegetable oils. The chemical name for testosterone cypionate is androst-4-en-3-one,17-(3-cyclopentyl-1oxopropoxy)-,
  (178)-. Its molecular formula is CvH400a, and the mole
- GA Genotype for the rs700518 Polymorphisms of the CYP19A1 Gene; AA Genotype for the rs700518 Polymorphism of the CYP19A1 Gene: All patients who qualify for the study will receive testosterone cypionate
  Testosterone Cypionate: DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Subjects were divided into the different genotypes for the rs700518 polymorphism of the CYP19A1 gene.
Arm/Group | GG Genotype for RS 700518 Polymorphism of the CYP19A1 Gene | GA Genotype for the rs700518 Polymorphisms of the CYP19A1 Gene | AA Genotype for the rs700518 Polymorphism of the CYP19A1 Gene
Number analyzed (Participants) | 15 | 44 | 25
percent change
  Lumbar spine | 3.69 (0.87) | 4.13 (0.52) | 3.82 (0.70)
  Total hip | 0.38 (0.93) | 0.93 (0.49) | 0.08 (0.66)
  Femoral neck | -1.09 (1.28) | 1.51 (0.69) | -1.25 (0.91)
Statistical Analysis 1: Comparison: GG Genotype for RS 700518 Polymorphism of the CYP19A1 Gene vs GA Genotype for the rs700518 Polymorphisms of the CYP19A1 Gene; Analysis by intention to treat with last value carry forward; Test type: Other; p < 0.05, ANOVA

2. Primary Outcome: Percent Change in Bone Mineral Density (BMD) According to the rs1062033 Polymorphism in the CYP19A1 Gene
Description: Percent change in bone mineral density from baseline to 18 months.
Time Frame: baseline to 18 months
Population: Analysis was by intention to treat with the last value carry forward. Those who had at least one follow-up from baseline were included in the analysis . The data of 82 subjects were available for analysis; 14 in the GG, 38 in the GC and 32 in the CC genotype.
Measure: Mean (Standard Deviation); unit: PERCENT CHANGE
Groups:
- GG Genotype of the rs1062033 Polymorphism in the CYP19A1 Gene: All patients who qualify for the study will receive testosterone cypionate
  Testosterone Cypionate: DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Subjects were divided into different genotypes of the rs1062033 polymorphism in the CYP19A1 gene
  Testosterone cypionate is a white or creamy white crystalline powder, odorless or nearly so and stable in air. It is insoluble in water, freely soluble in alcohol, chloroform, dioxane, ether, and soluble in vegetable oils. The chemical name for testosterone cypionate is androst-4-en-3-one,17-(3-cyclopentyl-1oxopropoxy)-,
  (178)-. Its molecular formula is CvH400a, and the mole
- GC Genotype of rs1062033 Polymorphism in the CYP19A1 Gene; CC Genotype for the rs1062033: All patients who qualify for the study will receive testosterone cypionate
  Testosterone Cypionate: DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Subjects were divided into different genotypes of the rs1062033 polymorphism in the CYP19A1 gene
Arm/Group | GG Genotype of the rs1062033 Polymorphism in the CYP19A1 Gene | GC Genotype of rs1062033 Polymorphism in the CYP19A1 Gene | CC Genotype for the rs1062033
Number analyzed (Participants) | 14 | 38 | 32
PERCENT CHANGE
  LUMBAR SPINE | 4.72 (0.91) | 2.85 (0.56) | 3.74 (0.63)
  FEMORAL NECK | -1.04 (1.31) | 0.64 (0.81) | 0.22 (0.96)
  TOTAL HIP | 0.33 (0.84) | 0.70 (0.50) | 0.64 (0.56)
Statistical Analysis 1: Comparison: GG Genotype of the rs1062033 Polymorphism in the CYP19A1 Gene vs GC Genotype of rs1062033 Polymorphism in the CYP19A1 Gene; Analysis by intention to treat with the last value carry forward; Test type: Other; p < 0.05, ANOVA

3. Secondary Outcome: Percent Change in Bone Mineral Density According to Body Mass Index (BMI)
Description: Percent changes in bone mineral density from baseline
Time Frame: baseline to 18 months
Population: Analysis was by intention to treat with the last value carry forward. Thirty subjects in BMI group 1, 31 in BMI group 2 and 23 subjects in BMI groups 3 have complete dataset available for analysis. There were a total 84 patients who were able to provide data for this outcome at 18 months.
Measure: Mean (Standard Error); unit: Percent change
Groups:
- BMI Group 1: All patients who qualify for the study will receive testosterone cypionate
  Testosterone Cypionate: DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Subjects were divided into different groups of BMI.
  Testosterone cypionate is a white or creamy white crystalline powder, odorless or nearly so and stable in air. It is insoluble in water, freely soluble in alcohol, chloroform, dioxane, ether, and soluble in vegetable oils. The chemical name for testosterone cypionate is androst-4-en-3-one,17-(3-cyclopentyl-1oxopropoxy)-,
  (178)-. Its molecular formula is CvH400a, and the mole
- BMI Group 2; BMI Group 3: All patients who qualify for the study will receive testosterone cypionate
  Testosterone Cypionate: DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Subjects were divided into different groups of BMI.
Arm/Group | BMI Group 1 | BMI Group 2 | BMI Group 3
Number analyzed (Participants) | 30 | 31 | 23
Percent change
  lumbar spine | 3.00 (0.97) | 4.90 (0.96) | 3.90 (1.24)
  Total hip | 0.14 (0.56) | 1.74 (0.55) | -0.27 (0.64)
  femoral neck | 0.71 (0.83) | -0.33 (0.86) | 0.16 (0.97)
Statistical Analysis 1: Comparison: BMI Group 1 vs BMI Group 2 vs BMI Group 3; Analysis by intention to treat with the last value carry forward; Test type: Other; p < 0.05, ANOVA

4. Secondary Outcome: Percent Change in Prostate-specific Antigen (PSA) According to the rs700518 Polymorphism of the CYP19A1 Gene
Description: Percent change in PSA from baseline to 18 months
Time Frame: From baseline to 18 months
Population: More participants came for their 6-month blood test than for other outcomes e.g. BMD. Since our analysis was intention to treat with the last value carry forward, there were more patients with evaluable PSA data at 18 months, as some patients who had PSA but had no BMD testing etc. who dropped out of the study were also included in the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- GG Genotype for the rs700518 Polymor[Hism of the CYP19A1 Gene: All patients who qualify for the study will receive testosterone cypionate
  Testosterone Cypionate: DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Subjects were divided into different genotypes for the rs700518 polymorphism of the CYP19A1 gene
  Testosterone cypionate is a white or creamy white crystalline powder, odorless or nearly so and stable in air. It is insoluble in water, freely soluble in alcohol, chloroform, dioxane, ether, and soluble in vegetable oils. The chemical name for testosterone cypionate is androst-4-en-3-one,17-(3-cyclopentyl-1oxopropoxy)-,
  (178)-. Its molecular formula is CvH400a, and the mole
- GA Genotype of the rs700518 Polymorphism in CYP19A1 Gen; AA Genotype for the rs700518 Polymorphism of the CYP19A1 Gene: All patients who qualify for the study will receive testosterone cypionate
  Testosterone Cypionate: DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Subjects were divided into different genotypes for the rs700518 polymorphism of the CYP19A1 gene
Arm/Group | GG Genotype for the rs700518 Polymor[Hism of the CYP19A1 Gene | GA Genotype of the rs700518 Polymorphism in CYP19A1 Gen | AA Genotype for the rs700518 Polymorphism of the CYP19A1 Gene
Number analyzed (Participants) | 17 | 46 | 26
percent change | 105.78 (167.93) | 58.52 (76.14) | 44.44 (59.92)
Statistical Analysis 1: Comparison: GG Genotype for the rs700518 Polymor[Hism of the CYP19A1 Gene vs GA Genotype of the rs700518 Polymorphism in CYP19A1 Gen; Analysis by intention to treat with the last value carry forward; Test type: Other; p < 0.05, ANOVA

5. Secondary Outcome: Percent Change in Prostate-specific Antigen (PSA) According to the rs1062033 Polymorphism of the CYP19A1 Gene
Description: Percent change in PSA from baseline at 18 months
Time Frame: from baseline to 18 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: precent change
Groups:
- CC Genotype for the rs1062033 Polymorphism in the CYP19A1 Gene: All patients who qualify for the study will receive testosterone cypionate
  Testosterone Cypionate: DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Subjects were divided into different genotypes of the rs1062033 polymorphism in the CYP19A1 gene
Arm/Group | GG Genotype of the rs1062033 Polymorphism in the CYP19A1 Gene | GC Genotype of rs1062033 Polymorphism in the CYP19A1 Gene | CC Genotype for the rs1062033 Polymorphism in the CYP19A1 Gene
Number analyzed (Participants) | 17 | 46 | 26
precent change | 85.15 (23.84) | 62.86 (15.74) | 52.93 (17.11)
Statistical Analysis 1: Comparison: GG Genotype of the rs1062033 Polymorphism in the CYP19A1 Gene vs GC Genotype of rs1062033 Polymorphism in the CYP19A1 Gene; Analysis by intention to treat with the last value carry forward; Test type: Other; p < 0.05, ANOVA

6. Secondary Outcome: Percent Change in Hematocrit According to the Genotype of the 700518 Polymorphism of the CYP19A1gene
Description: Percent change in hematocrit from baseline to 18 months
Time Frame: baseline to 18 months
Population: Analysis was by intention to treat with the last value carry forward. Those who had at least one follow-up from baseline were included in the analysis. The data of 85 subjects were available for analysis; 16 subjects in the GG, 43 in the GC and 26 subjects in the CC genotype.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- GG Genotype for the rs700518 Polymorphism of the CYP19A1 Gene: All patients who qualify for the study will receive testosterone cypionate
  Testosterone Cypionate: DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Subjects were divided according to the genotypes of rs700718 polymorphism of the CYP19A1 gene.
  Testosterone cypionate is a white or creamy white crystalline powder, odorless or nearly so and stable in air. It is insoluble in water, freely soluble in alcohol, chloroform, dioxane, ether, and soluble in vegetable oils. The chemical name for testosterone cypionate is androst-4-en-3-one,17-(3-cyclopentyl-1oxopropoxy)-,
  (178)-. Its molecular formula is CvH400a, and the mole
- GA Genotype for the rs700518 Polymorphism of the CYP19A1 Gene; AA Genotype for the rs700518 Polymorphism of the: All patients who qualify for the study will receive testosterone cypionate
  Testosterone Cypionate: DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Subjects were divided according to the genotypes of rs700718 polymorphism of the CYP19A1 gene.
Arm/Group | GG Genotype for the rs700518 Polymorphism of the CYP19A1 Gene | GA Genotype for the rs700518 Polymorphism of the CYP19A1 Gene | AA Genotype for the rs700518 Polymorphism of the
Number analyzed (Participants) | 16 | 43 | 26
Percent change | 11.32 (2.21) | 9.71 (1.35) | 9.41 (1.73)
Statistical Analysis 1: Comparison: GG Genotype for the rs700518 Polymorphism of the CYP19A1 Gene vs GA Genotype for the rs700518 Polymorphism of the CYP19A1 Gene; Analysis by intention to treat with the last value carry forward; Test type: Other; p < 0.05, ANOVA

7. Secondary Outcome: Percent Change in Hematocrit According to re1062033 Polymorphism of the CYP19A1 Gene
Description: Percent change in hematocrit from baseline to 18 months
Time Frame: Baseline to 18 months
Population: Analysis was by intention to treat with the last value carry forward. Those who had at least one follow-up from baseline were included in the analysis. The data of 85 subjects were available for analysis; 15 subjects in the GG, 37 in the GC and 33 subjects in the CC genotype.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- CC Genotype of rs1062033 Polymorphism in the CYP19A1 Gene: All patients who qualify for the study will receive testosterone cypionate
  Testosterone Cypionate: DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Subjects were divided into different genotypes of the rs1062033 polymorphism in the CYP19A1 gene.
Arm/Group | GG Genotype of the rs1062033 Polymorphism in the CYP19A1 Gene | GC Genotype of rs1062033 Polymorphism in the CYP19A1 Gene | CC Genotype of rs1062033 Polymorphism in the CYP19A1 Gene
Number analyzed (Participants) | 15 | 37 | 33
percent change | 11.56 (2.28) | 9.67 (1.45) | 9.46 (1.54)
Statistical Analysis 1: Comparison: GG Genotype of the rs1062033 Polymorphism in the CYP19A1 Gene vs GC Genotype of rs1062033 Polymorphism in the CYP19A1 Gene; Analysis by intention to treat with the last value carry forward; Test type: Other; p < 0.05, ANOVA

8. Secondary Outcome: Percent Change in Aromatase Gene Activity From the Buffy Coat According to the 700518 Polymorphism of the CYP19A1 Gene
Description: Percent change in gene expression from baseline to 18 months
Time Frame: Baseline to 6 months
Population: Gene expression studies were successful in 27 samples; 6 in the GG, 17 in the GA and 4 in the AA genotype.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | GG Genotype for the rs700518 Polymorphism in the cYP19A1 Gene | GA Genoypr for the rs700518 Polymorphism of the CYP19A1 Gene | AA Genotype for the rs700518 Polymorphism of the CYP19A1 Gene
Number analyzed (Participants) | 6 | 17 | 4
percent change | 25.0 (120.0) | 65.25 (71.29) | 113.33 (146.97)

9. Secondary Outcome: Percent Change in Bone Turnover Markers According to the rs700518 Polymorphism of the CYP19A1 Gene
Description: Percent change in bone turnover from baseline to 18 months.
Time Frame: Baseline to 18 months
Population: Analysis was by intention to treat with the last value carry forward. Those who had at least one follow-up from baseline were included in the analysis. The data of 79 subjects were analyzed; 15 in the GG, 43 in the GA and 21 in the AA genotype.
Measure: Mean (Standard Deviation); unit: perecent change
Groups:
- GG Genotype for RS 700518 of the CYP19A1 Gene: All patients who qualify for the study will receive testosterone cypionate
  Testosterone Cypionate: DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Subjects were divided into the different genotypes for the rs700518 polymorphism of the CYP19A1 gene.
  Testosterone cypionate is a white or creamy white crystalline powder, odorless or nearly so and stable in air. It is insoluble in water, freely soluble in alcohol, chloroform, dioxane, ether, and soluble in vegetable oils. The chemical name for testosterone cypionate is androst-4-en-3-one,17-(3-cyclopentyl-1oxopropoxy)-,
  (178)-. Its molecular formula is CvH400a, and the mole
- GA Genotype for the rs700518 Polymorphism of the CYP19A1 Gene; AA Genotype for the rs700518 Polymorphism of the CYP19A1 Gene: All patients who qualify for the study will receive testosterone cypionate
  Testosterone Cypionate: DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Subjects were divided into the different genotypes for the rs700518 polymorphism of the CYP19A1 gene.
Arm/Group | GG Genotype for RS 700518 of the CYP19A1 Gene | GA Genotype for the rs700518 Polymorphism of the CYP19A1 Gene | AA Genotype for the rs700518 Polymorphism of the CYP19A1 Gene
Number analyzed (Participants) | 15 | 43 | 21
perecent change
  C-teloepetide | 41.47 (16.33) | 3.35 (9.64) | -9.75 (13.80)
  Osteocalcin | 12.40 (133.13) | -31.22 (148.00) | -7.27 (112.06)
Statistical Analysis 1: Comparison: GG Genotype for RS 700518 of the CYP19A1 Gene vs GA Genotype for the rs700518 Polymorphism of the CYP19A1 Gene; Analysis was by intention to treat with the last value carry forward. Those who had at least one follow-up from baseline and with acceptable assay coefficient of variability were included in the analysis. The data of 79 subjects were analyzed; 15 in the GG, 43 in the GA and 21 in the AA genotype; Test type: Other; p < 0.05, ANOVA

10. Secondary Outcome: Percent Change in Bone Turnover Markers According to the rs1062033 Polymorphism of the CYP19A1 Gene
Description: Percent change in bone turnover markers
Time Frame: Baseline to 18 months
Population: Analysis was by intention to treat with the last value carry forward. Those who had at least one follow-up from baseline were included in the analysis. The data of 79 subjects with acceptable assay coefficient of variability were available for analysis; 15 subjects in the GG, 37 in the GC and 27 in the CC genotype.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- GG Genotype for the rs1062033 Polymorphism of the CYP19A1 Gene: All patients who qualify for the study will receive testosterone cypionate
  Testosterone Cypionate: DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Subjects were divided according to the genotypes of rs1062033 polymorphism of the CYP19A1 gene.
  Testosterone cypionate is a white or creamy white crystalline powder, odorless or nearly so and stable in air. It is insoluble in water, freely soluble in alcohol, chloroform, dioxane, ether, and soluble in vegetable oils. The chemical name for testosterone cypionate is androst-4-en-3-one,17-(3-cyclopentyl-1oxopropoxy)-,
  (178)-. Its molecular formula is CvH400a, and the mole
- GC Genotype for the rs1062033 Polymorphism of the; GG Genotype for the rs1062033 Polymorphism in the CYP19A1 Gene: All patients who qualify for the study will receive testosterone cypionate
  Testosterone Cypionate: DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Subjects were divided according to the genotypes of 1062033 polymorphism of the CYP19A1 gene.
Arm/Group | GG Genotype for the rs1062033 Polymorphism of the CYP19A1 Gene | GC Genotype for the rs1062033 Polymorphism of the | GG Genotype for the rs1062033 Polymorphism in the CYP19A1 Gene
Number analyzed (Participants) | 15 | 37 | 27
Percent change
  C-telopeptide | 48.96 (98.42) | 5.89 (48.82) | -14.49 (51.05)
  Osteocalcin | 33.59 (118.59) | -20.59 (128.37) | -26.96 (144.48)
Statistical Analysis 1: Comparison: GG Genotype for the rs1062033 Polymorphism of the CYP19A1 Gene vs GC Genotype for the rs1062033 Polymorphism of the; Analysis by intention to treat with the last value carry forward; Test type: Other; p < 0.05, ANOVA

11. Secondary Outcome: Percent Change in Bone Mineral Density According the Presence of Diabetes Mellitus
Description: Percent change in bone mineral density from baseline to 18 months
Time Frame: Baseline to 18 months
Population: Analysis was by intention to treat with the last value carry forward. Thirty-nine subjects with diabetes mellitus group and 45 without diabetes mellitus have complete dataset available for analysis.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Subjects With Diabetes Mellitus: All patients who qualify for the study will receive testosterone cypionate
  Testosterone Cypionate: DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Subjects were divided into those with and without diabetes mellitus.
  Testosterone cypionate is a white or creamy white crystalline powder, odorless or nearly so and stable in air. It is insoluble in water, freely soluble in alcohol, chloroform, dioxane, ether, and soluble in vegetable oils. The chemical name for testosterone cypionate is androst-4-en-3-one,17-(3-cyclopentyl-1oxopropoxy)-,
  (178)-. Its molecular formula is CvH400a, and the mole
- Subjects Without Diabetes Mellitus: All patients who qualify for the study will receive testosterone cypionate
  Testosterone Cypionate: DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Subjects were divided into those with and without diabetes mellitus.
Arm/Group | Subjects With Diabetes Mellitus | Subjects Without Diabetes Mellitus
Number analyzed (Participants) | 39 | 45
Percent change
  LUMBAR SPINE | 4.05 (0.60) | 3.28 (0.51)
  TOTAL HIP | 1.81 (0.61) | 0.53 (0.49)
  FEMORAL NECK | 1.63 (0.95) | -0.55 (0.79)
Statistical Analysis 1: Comparison: Subjects With Diabetes Mellitus vs Subjects Without Diabetes Mellitus; Analysis by intention to treat with the last value carry forward; Test type: Other; p < 0.05, ANOVA

12. Secondary Outcome: Percent Change in Bone Turnover Markers According the Presence of Diabetes Mellitus
Description: Percent change in bone turnover markers from baseline to 18 months.
Time Frame: Baseline to 18 months
Population: Analysis was by intention to treat with the last value carry forward. Thirty-seven subjects with diabetes mellitus group and 41 without diabetes mellitus have complete dataset available for analysis.
Measure: Mean (Standard Error); unit: Percentage Changes
Arm/Group | Subjects With Diabetes Mellitus | Subjects Without Diabetes Mellitus
Number analyzed (Participants) | 37 | 41
Percentage Changes
  C-telopeptide | 73.55 (22.88) | 2.05 (16.22)
  Osteocalcin | 20.54 (15.64) | -6.62 (10.54)
Statistical Analysis 1: Comparison: Subjects With Diabetes Mellitus vs Subjects Without Diabetes Mellitus; Analysis by intention to treat with the last value carry forward; Test type: Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 18 months
Groups:
- Arm 1: Testosterone Cypionate: All patients who qualify for the study will receive testosterone cypionate
  Testosterone Cypionate: DEPo-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble 17 (beta)-cyclopentylpropionate ester of the androgenic hormone testosterone.
  Testosterone cypionate is a white or creamy white crystalline powder, odorless or nearly so and stable in air. It is insoluble in water, freely soluble in alcohol, chloroform, dioxane, ether, and soluble in vegetable oils. The chemical name for testosterone cypionate is androst-4-en-3-one,17-(3-cyclopentyl-1oxopropoxy)-,
  (178)-. Its molecular formula is CvH400a, and the mole
Arm/Group | Arm 1: Testosterone Cypionate
All-Cause Mortality (participants affected / at risk) | 0/105
Serious Adverse Events (participants affected / at risk) | 18/105
Other Adverse Events (participants affected / at risk) | 51/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Testosterone Cypionate (N=105)
stroke (Nervous system disorders) | 2
abscess (Infections and infestations) | 1
appendicitis (Gastrointestinal disorders) | 1
GI tract perforation (Gastrointestinal disorders) | 1
infection of an appendectomy wound (Infections and infestations) | 1
pyschiatric ilness (Psychiatric disorders) | 4 — suicidal ideation
knee arthroscopy (Musculoskeletal and connective tissue disorders) | 1
knee replacement surgery (Musculoskeletal and connective tissue disorders) | 1
coronary stent (Cardiac disorders) | 2
atypical chest pain (Cardiac disorders) | 1
new-onset atrial fibrillation (Cardiac disorders) | 1
myocardial infarction (Cardiac disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Testosterone Cypionate (N=105)
Congestive heart failure (Cardiac disorders) | 1
appendicitis (Gastrointestinal disorders) | 1
diverticulitis (Gastrointestinal disorders) | 2
heartburn (Gastrointestinal disorders) | 1
gallstones (Hepatobiliary disorders) | 1
infected appendectomy wound (Gastrointestinal disorders) | 1
infected spider bite (Infections and infestations) | 1
shingles (Infections and infestations) | 1
cellulitis (Infections and infestations) | 1
high hematocrit (Blood and lymphatic system disorders) | 9
hemochromatosis (Blood and lymphatic system disorders) | 1
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
lung carcinoma (Respiratory, thoracic and mediastinal disorders) | 1
priapism (Reproductive system and breast disorders) | 1
mastitis (Reproductive system and breast disorders) | 1
prostate enlargement (Renal and urinary disorders) | 1
alopecia (Skin and subcutaneous tissue disorders) | 1
acne (Skin and subcutaneous tissue disorders) | 1
laceration (Skin and subcutaneous tissue disorders) | 3
mood swings (Psychiatric disorders) | 1
irritability (Psychiatric disorders) | 1
depression (Psychiatric disorders) | 1
headache (Nervous system disorders) | 1
ingrown toenail (Musculoskeletal and connective tissue disorders) | 1
heel pain (Musculoskeletal and connective tissue disorders) | 1
arthroplasty (Musculoskeletal and connective tissue disorders) | 3
foot pain (Musculoskeletal and connective tissue disorders) | 1
vertebral fracture (Musculoskeletal and connective tissue disorders) | 1
osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
excision of bone spur (Musculoskeletal and connective tissue disorders) | 2
knee replacement (Musculoskeletal and connective tissue disorders) | 1
sleep apnea (General disorders) | 1
back pain (Injury, poisoning and procedural complications) | 1
retinal injury (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes